CLINICAL TRIAL: NCT05688540
Title: Efficiency of Electronic Multimedia Intervention on Quality of Life, Psychological Adjustment and Depression in Patients With the Cardiac Implantable Electronic Device
Brief Title: Efficiency of Electronic Multimedia Intervention With the Cardiac Implantable Electronic Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Miao Yen Chen, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18MMHIS006e
Record Dates: First submitted 2023-01-07; First posted 2023-01-18 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Implantable Electronic Device
Keywords: cardiac implantable electronic device; quality of life; electronic multimedia; psychological adjustment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e book (Experimental): a multi-media model through e-book for preoperative care of CIED intervention.
  Interventions: Other: e book
- traditional education booklet (Experimental): traditional education booklet of CIED intervention.
  Interventions: Other: traditional education booklet

INTERVENTIONS:
Other: e book — e book
  Arms: e book
Other: traditional education booklet — traditional education booklet
  Arms: traditional education booklet

SUMMARY:
In this study, we aim to design a multi-media model through e-book for preoperative care of CIED intervention, which can enhance the knowledges of patients, reducing the stresses and uncertainties before the intervention. Therefore, patient may reduce the psychological internalization after CIED intervention, also needs to track the impact of emotional depression, psychological adaption and life quality status.

DETAILED DESCRIPTION:
Arrhythmia is defined an abnormality in the heart transmission system related to heartbeat or heart rhythm problem (Li et al., 2017). Most of arrhythmia could diagnosed and treated effectively, including medication, cardiac implantable electronic device (CIED) and operation. Many patients have uncertainty about the implantation process, the results and possible complications after CIED, the lack of understanding about further progress of their disease, the change of lifestyle and the accident of electronic shock. Those causes are the physical and mental negative impacts on patient which makes anxiety or depressed and turn affects the quality of life.

At present, there are few clinical models for CIED utilizing electronic multi-media in Taiwan. The use of multi-media models may integrate clinical care and health education for helping patients to learn disease and care, also through vivid video and multi-media, we may make a clear education of disease causes, treatment and relevant care knowledges which are alleviate the uncertainty factors from patients (Hsueh et al., 2016). Therefore, the more overall understanding before CIED intervention, the more helpful to quality of living and psychological adjustment of the patient.

In this study, we aim to design a multi-media model through e-book for preoperative care of CIED intervention, which can enhance the knowledges of patients, reducing the stresses and uncertainties before the intervention. Therefore, patient may reduce the psychological internalization after CIED intervention, also needs to track the impact of emotional depression, psychological adaption and life quality status.

keywords：Cardiac Implantable Electronic Device、arrhythmia、electronic multimedia、quality of life、psychological adjustment、depression

ELIGIBILITY:
Inclusion Criteria:

1. Actual age > 20 years-old adults.
2. Patients are willing to participate in this research.
3. Conscious clear, sanity, and be able to communicate with others in Mandarin or Taiwanese languages.
4. Be able to operate mobile electronic device, such as mobile phone, iPAD or laptop; Families and healthcare provider allows to assist.

Exclusion Criteria:

1. TDS > score 19 (Severely depressed patient)
2. Patient of terminal stage cancer.
3. Patient with delirium during hospitalization.

Ages: 20 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF(TW) | 20mins
  28 questions totally with four parts, including physical, mental, social-behavior related and environment aspects. The more score they get, means more quality of life they obtained.
Chinese 14-item PSS | 10mins
  14 questions totally for measuring the stress of patient in a month.
Taiwan Depression Scale | 10mins
  18 questions totally for testing how level of anxiety and depress of patient. The element of this scale are mental aspect, self-thought aspect and physical aspect.

CONTACTS AND LOCATIONS:
Overall Officials: Yen Chen CHEN, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasi M, Negarandeh R, Norouzadeh R, Shojae Mogadam AR. The Challenges of Living With an Implantable Cardioverter Defibrillator: A Qualitative Study. Iran Red Crescent Med J. 2016 Jun 22;18(10):e25158. doi: 10.5812/ircmj.25158. eCollection 2016 Oct. PMID 28180011